CLINICAL TRIAL: NCT00119769
Title: The Effect of Low-Dose Human Growth Hormone Therapy in HIV Infected Patients on Highly Active Antiretroviral Therapy (HAART)
Brief Title: The Effect of Low-Dose Human Growth Hormone Therapy in HIV Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Ove Andersen, Clinical Research Center, Copenhagen University Hospital Hvidovre, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KFE001
Record Dates: First submitted 2005-07-07; First posted 2005-07-14 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: HIV Infections; Lipodystrophy
Keywords: HIV; immune stimulation; lipodystrophy; growth hormone; recombinant growth hormone; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Lipodystrophy | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Active Comparator)
  Interventions: Drug: Genotropin (human recombinant Growth hormone)

INTERVENTIONS:
Drug: Placebo — Placebo, 0.7 mg/day injected subcutaneously
  Arms: 1
Drug: Genotropin (human recombinant Growth hormone) — Genotropin, 0.7 mg/day injected subcutaneously
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the effect of low-dose human growth hormone therapy on immune status and fat morphology.

DETAILED DESCRIPTION:
Following the introduction of highly active antiretroviral therapy (HAART) in the mid-nineties, the improvement in the clinical course of HIV has lead to a dramatic reduction in morbidity and mortality. However, a growing concern has been the emergence of an increasing number of drug therapy failure, mainly caused by rebounding virus. This effect in turn is prompted respectively by developing resistance and failing compliance mainly due to early or late adverse reactions. These adverse reactions mainly consists of a number of metabolic and morphologic changes, known as HIV associated lipodystrophy syndrome (HALS) and affects approximately 40 % of HIV infected patients on HAART. HALS is characterized by lipoatrophy on extremities, gluteal and facial regions combined with intraabdominal lipoaccumulation, "buffalo hump" and lipomas.

Thus, despite progress in the development of new drugs with new targets and resistance profiles the need for agents with immune modulating properties is evident, both as a way to overcome the problems of resistance and hopefully modify treatment regimens in order to reduce the exposure to late adverse reactions caused by HAART. A number of studies have addressed the problems of modulating the immune response during HIV infection. Results are promising but a major obstacle seems to be adverse effects. In the pre-HAART era high dose human growth hormone (hGH) therapy has been used for HIV wasting and in the HAART era the impact on fat distribution in HIV infected patients have been investigated based on the lipolytic properties of hGH. However high dosage of hGH has been associated with severe adverse effects limiting the usefulness in daily clinical practice. One recent study demonstrated increments in thymic mass and a rise in the number of circulating naïve CD4 T cells upon treatment with high dose hGH. Our group has conducted a 60 week pilot study with daily injection of 0.7 mg genotropin, demonstrating an immune stimulating effect as well as an increased limb fat/truncal fat ratio, without metabolic and clinically recognizable side effects. Based on these findings we plan to perform a randomized, double blind, prospective, interventional study including 50 HIV infected patients on HAART, investigating the effect of low dose hGH on immune status and fat distribution.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Caucasian race
* Age >21 years, <60 years
* HIV-1 infection
* HAART treated > 12 months
* HIV-RNA < 100 copies/ml
* CD4 count > 200
* Fasting plasma glucose < 6.1 mM
* Stable weight

Exclusion Criteria:

* BMI > 28 kg/m2 and BMI < 18.5 kg/m2
* Wasting or AIDS defining disease
* Severe chronic diseases other than HIV
* Cancer, previous transplantation
* Previous AMI
* Diabetes
* Hormonal substitution therapy
* Lipid lowering or antidiabetic therapy within 3 months
* Abuse of narcotics or alcohol
* Major psychiatric disorders
* Adverse reactions towards Genotropin
* Calcium-ion < 1.15 or > 1.35 mM
* D-vitamin < 19 nM
* TSH < 0.1 or > 10 mIU/l

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2005-02; Primary Completion 2007-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Impact of hGH 0.7 mg/day on number of mature and naïve CD4 cells in HIV patients at 9 months | 9 months

SECONDARY OUTCOMES:
Impact of hGH 0.7 mg/day at 9 months on thymic size | 9 months
Impact of hGH 0.7 mg/day at 9 months on fat distribution as measured with CT and DEXA scans | 9 months
Impact of hGH 0.7 mg/day at 9 months on glucose metabolism i.e.glucose tolerance, insulin sensitivity and beta cell function as measured by OGTT | 9 months
Impact of hGH 0.7 mg/day at 9 months on insulin sensitivity as measured by hyperinsulinaemic euglycaemic clamp | 9 months
Impact of hGH 0.7 mg/day at 9 months on lipid profile | 9 months
Impact of hGH 0.7 mg/day at 9 months on quality of life and adherence to HAART | 9 months
Impact of hGH 0.7 mg/day at 9 months on cytokines | 9 months
Impact of hGH 0.7 mg/day at 9 months on safety parameters | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte R Hansen, MD, Principal Investigator
Locations (1):
- Clinical Research Unit, Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Background] Andersen O, Haugaard SB, Hansen BR, Orskov H, Andersen UB, Madsbad S, Iversen J, Flyvbjerg A. Different growth hormone sensitivity of target tissues and growth hormone response to glucose in HIV-infected patients with and without lipodystrophy. Scand J Infect Dis. 2004;36(11-12):832-9. doi: 10.1080/00365540410021162. PMID 15764170
- [Background] Haugaard SB, Andersen O, Dela F, Holst JJ, Storgaard H, Fenger M, Iversen J, Madsbad S. Defective glucose and lipid metabolism in human immunodeficiency virus-infected patients with lipodystrophy involve liver, muscle tissue and pancreatic beta-cells. Eur J Endocrinol. 2005 Jan;152(1):103-12. doi: 10.1530/eje.1.01835. PMID 15762193
- [Background] Haugaard SB, Andersen O, Volund A, Hansen BR, Iversen J, Andersen UB, Nielsen JO, Madsbad S. Beta-cell dysfunction and low insulin clearance in insulin-resistant human immunodeficiency virus (HIV)-infected patients with lipodystrophy. Clin Endocrinol (Oxf). 2005 Mar;62(3):354-61. doi: 10.1111/j.1365-2265.2005.02223.x. PMID 15730419
- [Background] Haugaard SB, Andersen O, Hansen BR, Andersen UB, Volund A, Iversen J, Nielsen JO, Madsbad S. In nondiabetic, human immunodeficiency virus-infected patients with lipodystrophy, hepatic insulin extraction and posthepatic insulin clearance rate are decreased in proportion to insulin resistance. Metabolism. 2005 Feb;54(2):171-9. doi: 10.1016/j.metabol.2004.08.009. PMID 15690310
- [Background] Haugaard SB, Andersen O, Hansen BR, Orskov H, Andersen UB, Madsbad S, Iversen J, Flyvbjerg A. Insulin-like growth factors, insulin-like growth factor-binding proteins, insulin-like growth factor-binding protein-3 protease, and growth hormone-binding protein in lipodystrophic human immunodeficiency virus-infected patients. Metabolism. 2004 Dec;53(12):1565-73. doi: 10.1016/j.metabol.2004.06.025. PMID 15562401
- [Background] Andersen O, Haugaard SB, Flyvbjerg A, Andersen UB, Orskov H, Madsbad S, Nielsen JO, Iversen J. Low-dose growth hormone and human immunodeficiency virus-associated lipodystrophy syndrome: a pilot study. Eur J Clin Invest. 2004 Aug;34(8):561-8. doi: 10.1111/j.1365-2362.2004.01380.x. PMID 15305891